CLINICAL TRIAL: NCT05502003
Title: Effect Of High Intensity Interval Upper Extremity Training On Biochemistry Parameters And Disease Symptoms In Patients With Fibromyalgia
Brief Title: The Effect of Telerehabilitation on Symptoms in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Selin Akıl Ağdere, Physiotherapist, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aerobic exercise
Record Dates: First submitted 2022-08-10; First posted 2022-08-16 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; high intensity interval training; telerehabilitation; tryptophan
MeSH Terms: conditions — Fibromyalgia | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Interval Training (Experimental): With the arm ergometer given to the participants, a telerehabilitation-based upper extremity aerobic exercise program will be applied. Maximum Heart Rate (MHR) will be determined by the formula '220-age', and exercise intensity will be calculated, and exercise will begin with a 5 minute warm-up. Cycle will be created with 4 min MHR (80-95%) high intensity and 3 min MHR (70%) active recovery and exercise will be terminated with 5 min cool down. A total of 35 minutes of exercise program will be given.
  Interventions: Other: High Intensity Interval Training
- Moderate Exercise Training (Active Comparator): An upper extremity exercise program with telerehabilitation (Zoom/videoconference) will be applied to the moderate-intensity exercise group. Maximum heart rate (MHR) will be determined by the formula 220-Age. A total of 55 minutes of moderate exercise training will be given at 65-70% of MHR, with five minutes of warm-up and cool-down.
  Interventions: Other: Moderate Exercise Training
- Control (No Intervention): No aerobic exercise program will be applied to this group.

INTERVENTIONS:
Other: High Intensity Interval Training — Telerehabilitation-based high-intensity exercise training will be applied to the participants for 6 weeks, 3 times a week for 35 minutes, under the control of a physiotherapist.
  Arms: High Intensity Interval Training
Other: Moderate Exercise Training — The participants will be given telerehabilitation-based moderate exercise training under the control of a physiotherapist for 55 minutes, 3 times a week for 6 weeks.
  Arms: Moderate Exercise Training

SUMMARY:
The aim of this study is to evaluate the effect of telerehabilitation-based high-intensity interval upper extremity exercise training on biochemistry parameters and disease symptoms in fibromyalgia patients. It has been reported that substances such as serotonin and tryptophan are found at abnormal levels in the serotonergic system in patients with fibromyalgia, and symptoms such as depression, pain, and fatigue related to the disease may be associated with this condition. In the literature, there are studies conducted in other disease groups showing that aerobic exercise regulates tryptophan and serotonin levels and can produce positive results regarding these symptoms. This study was planned to evaluate the effect of high-intensity interval exercise training, which is an aerobic exercise form, whose benefits are frequently mentioned in recent publications, on both blood parameters and symptoms in fibromyalgia patients.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic musculoskeletal disease of unknown etiology accompanied by symptoms such as pain, hyperalgesia, sleep disorders, fatigue and mood disorders. It has been suggested that a defect in the serotonergic system is involved in the pathophysiology of the disease. The serotonergic system has been associated with many symptoms such as anxiety, depression, sleep problems, fatigue and pain. In studies on fibromyalgia, it was reported that plasma tryptophan and serotonin levels decreased in this patient group and that serotonin levels were abnormal in the endogenous pain blocking pathways. Although conflicting results have been reported, it was stated that vitamin D levels were also low in this patient group. Aerobic exercise makes muscles use branched-chain amino acids, reducing the amount of amino acids that compete with tryptophan and increasing the chance of tryptophan to cross the blood-brain barrier. Therefore, it has the potential to increase serotonin in the brain. In particular, aerobic exercise appears to modulate hormone, neurotrophin and neurotransmitter levels, depending on factors such as genes, age and hormonal status. On the other hand, it is reported that some types of exercise increase the production of free radicals and cause oxidative stress. It has been suggested that oxidative stress may be associated with pain, which is one of the main symptoms in fibromyalgia patients by affecting nociceptors. Studies have shown that when aerobic exercises are applied regularly for a long time, lipid peroxidation level, which is an indicator of oxidative stress, decreases and antioxidant enzyme activity increases. Regularly applied aerobic exercise programs have been reported as a suitable form of exercise for this patient group. Recent studies have focused on high-intensity interval training. This type of exercise; It is performed as successive short and intermittent sessions of high-intensity activity with periods of low intensity or rest. High-intensity interval training are shorter than moderate aerobic workouts and produce the same or more positive effects than moderate exercise. It is also reported that high-intensity interval training application improves oxidative capacity, antioxidant defense and endothelial functions. Telerehabilitation practices refer to the use of telematics procedures using telephone, video and computer technologies instead of traditional face-to-face approaches. The therapist ensures that patient communication and follow-up are maintained by maintaining social distance. It has been stated in studies that telerehabilitation can be used to increase the quality of life, to provide socialization and to treat pain in patients with fibromyalgia. This study was designed to evaluate the effectiveness of high-intensity interval training upper extremity exercise training, which is a form of aerobic exercise, on these parameters, associated symptoms and oxidative stress markers in fibromyalgia patients with negative effects on serotonin, tryptophan, vitamin D and related parameters.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with fibromyalgia according to the American College of Rheumatology 2016 criteria.
* Participants between the ages of 18-65
* Participants who do not use a drug that will affect the treatment results
* Participants who volunteer

Exclusion Criteria:

* Infection
* Fever
* Any known advanced-stage pathology associated with the locomotor system that contraindicates physical activity.
* Cardiopulmonary problem
* Presence of autoimmune disease
* Pregnancy
* Malignancy
* Severe psychiatric problem
* Neurological disorder
* Epilepsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Assessment of serum free tryptophan | 6 weeks
  Blood will be drawn from the participants in the morning. Centrifugation will be performed and the blood taken will be frozen.The analysis will be completed by following the manufacturer's instructions of the appropriate kits.
Assessment of 5-Hydroxyindolacetic Acid | 6 weeks
  Blood will be drawn from the participants in the morning. Centrifugation will be performed and the blood taken will be frozen.The analysis will be completed by following the manufacturer's instructions of the appropriate kits.
Assessment of Superoxide dismutase | 6 weeks
  Superoxide dismutase is the most important enzymatic antioxidants that prevent the initiation of lipid peroxidation. Blood will be drawn from the participants in the morning. Centrifugation will be performed and the blood taken will be frozen. The analysis will be completed by following the manufacturer's instructions of the appropriate kits.
Assessment of Glutathione Peroxidase | 6 weeks
  Glutathione Peroxidase is the most important enzymatic antioxidants that prevent the initiation of lipid peroxidation. Blood will be drawn from the participants in the morning. Centrifugation will be performed and the blood taken will be frozen. The analysis will be completed by following the manufacturer's instructions of the appropriate kits.
Assessment of Malondialdehyde | 6 weeks
  Blood will be drawn from the participants in the morning. Centrifugation will be performed and the blood taken will be frozen. The analysis will be completed by following the manufacturer's instructions of the appropriate kits.
Assessment of Myeloperoxidase | 6 weeks
  Blood will be drawn from the participants in the morning. Centrifugation will be performed and the blood taken will be frozen. The analysis will be completed by following the manufacturer's instructions of the appropriate kits.
Assessment of 25-hydroxy vitamin D | 6 weeks
  Blood will be drawn from the participants in the morning. Centrifugation will be performed and the blood taken will be frozen. The analysis will be completed by following the manufacturer's instructions of the appropriate kits.

SECONDARY OUTCOMES:
Pressure Pain Threshold Assessment | 6 weeks
  Pressure pain threshold assessment will be done with an algometer.
Evaluation of Grip Strength | 6 weeks
  Grip strength will be evaluated with a dynamometer (Hydraulic hand dynamometer).
Evaluation of Fatigue | 6 weeks
  Fatigue will be evaluated with Fatigue Severity Scale. Each item of the scale, which consists of 9 items that patients can apply on their own, is scored between 1 and 7 (1 = strongly disagree, 7 = completely agree) and the total score is calculated by taking the average of 9 items. The lower the total score, the less fatigue.
Evaluation of Depression and Anxiety | 6 weeks
  Depression and anxiety will be evaluated with Hospital Anxiety and Depression Scale. Each item of the 14-item scale is scored between 0 and 3. For anxiety and depression values, 0-7 points are considered normal, 8-10 points are borderline, and 11 points and above are considered abnormal.
Evaluation of Quality of Sleep | 6 weeks
  Quality of Sleep will be evaluated with Pittsburgh Sleep Quality Index. The total score is between 0-21. A high total score indicates poor sleep quality.
Evaluation of Functional Status Assessment | 6 weeks
  Functional Status Assessment will be evaluated with The Revised Fibromyalgia Impact Questionnaire. A high score indicates that the disease affects the person more.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Bakırköy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Bakırköy, Turkey (Türkiye)

REFERENCES:
- [Background] Schwarz MJ, Offenbaecher M, Neumeister A, Ackenheil M. Experimental evaluation of an altered tryptophan metabolism in fibromyalgia. Adv Exp Med Biol. 2003;527:265-75. doi: 10.1007/978-1-4615-0135-0_30. PMID 15206740
- [Background] Siracusa R, Paola RD, Cuzzocrea S, Impellizzeri D. Fibromyalgia: Pathogenesis, Mechanisms, Diagnosis and Treatment Options Update. Int J Mol Sci. 2021 Apr 9;22(8):3891. doi: 10.3390/ijms22083891. PMID 33918736